CLINICAL TRIAL: NCT05563844
Title: An Open-label, Multi-center Phase II Clinical Study on the Efficacy and Safety of Purinostat Mesylate for Injection in the Treatment of Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Study of Purinostat Mesylate for Injection in the Treatment of Relapsed or Refractory Diffuse Large B-cell Lymphoma (R/R DLBCL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZLPM-001-1.0
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B Cell Lymphoma，DLBCL
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purinostat Mesylate for Injection 8.4mg/m^2 (Experimental): The medication is administered once via intravenous infusion on days 1, 4, 8, and 11 of each 21-day treatment cycle.
  Interventions: Drug: PM 8.4 mg/m^2
- Purinostat Mesylate for Injection 11.2mg/m^2 (Experimental): The medication is administered once via intravenous infusion on days 1, 4, 8, and 11 of each 21-day treatment cycle.
  Interventions: Drug: PM 11.2 mg/m^2

INTERVENTIONS:
Drug: PM 8.4 mg/m^2 — The medication is administered once via intravenous infusion on days 1, 4, 8, and 11 of each 21-day treatment cycle. A total of 6 cycles are planned, with tumor response assessments performed every 2 cycles during the treatment period.
  Arms: Purinostat Mesylate for Injection 8.4mg/m^2
Drug: PM 11.2 mg/m^2 — The medication is administered once via intravenous infusion on days 1, 4, 8, and 11 of each 21-day treatment cycle. A total of 6 cycles are planned, with tumor response assessments performed every 2 cycles during the treatment period.
  Arms: Purinostat Mesylate for Injection 11.2mg/m^2

SUMMARY:
Purinostat mesylate for injection (PM) was the novel and highly potent Class Ia and IIb HDAC selective inhibitor. The results of regular blood sampling analysis of the mouse B-cell lymphoma model induced by ighmyc transgenic mice showed that the treatment of PM in each group reduced the proportion of peripheral blood tumor cells in mice. Therefore, PM has the potential to treat diffuse large B cell lymphoma.

Compared with the blank control group, the body weight of the tumor-bearing animals in each dose of PM group did not decrease significantly during the treatment process, and the animals were in good condition during the whole experiment, indicating that the PM is efficacious and safe.

Main purpose:

To further explore the safe and effective dose of purinostat mesylate for injection in the treatment of relapsed or refractory diffuse large B-cell lymphoma.

To evaluate the objective response rate (ORR) of purinostat mesylate for injection in the treatment of relapsed or refractory diffuse large B-cell lymphoma.

Secondary purpose:

To evaluate the time to tumor response (TTR), duration of response (DOR), disease control rate (DCR), and progression-free survival (PFS) in the treatment of relapsed or refractory diffuse large B-cell lymphoma with purinostat mesylate for injection ), overall survival (OS).

Assessing the safety and tolerability of purinostat mesylate for injection in the treatment of relapsed or refractory diffuse large B-cell lymphoma.

Exploratory purpose:

To explore the biomarkers related to the efficacy of purinostat mesylate for injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, both males and females are eligible;
2. Histologically confirmed diffuse large B-cell lymphoma (DLBCL) by tissue biopsy (including primary DLBCL and transformed DLBCL from indolent lymphoma; patients with relapse after more than one year require a repeat tissue biopsy to confirm the pathological diagnosis), and must be relapsed/refractory, specifically defined as: DLBCL patients who have received no more than 5 lines of prior systemic therapy. Relapse includes: 1) relapse occurring more than 6 months after the completion of second-line therapy; 2) relapse occurring more than 3 months after sequential hematopoietic stem cell transplantation following second-line therapy. Refractory includes: 1) primary refractory to first-line standard therapy (i.e., no response to treatment or relapse within 6 months after treatment completion); 2) relapse within 6 months after second-line therapy or failure to achieve partial response (PR) after 2 or more cycles of second-line therapy, or progression during second-line therapy (no specific cycle requirement for refractory patients). Prior treatment must include anti-CD20 monoclonal antibody (unless contraindicated) and anthracycline-based chemotherapy (unless anthracycline is contraindicated). Anti-CD20 monoclonal antibody monotherapy for consolidation or induction does not count as a separate line of therapy. Prior stem cell transplantation is allowed; standalone autologous stem cell transplantation does not count as a line of therapy, as induction, consolidation, stem cell collection, conditioning regimen, and transplantation ± maintenance therapy are considered one line of therapy.
3. Presence of measurable lesions, defined as: lymph node lesions with the longest diameter > 15 mm or extranodal lesions with the longest diameter > 10 mm as measured by contrast-enhanced CT, MRI, or PET-CT; willingness to undergo bone marrow aspiration cytology and/or biopsy for efficacy evaluation if required.
4. Prior to the first dose of study treatment, the following intervals must be observed: ≥ 4 weeks since the last systemic radiotherapy; ≥ 2 weeks since local radiotherapy or radiotherapy for bone metastases; no radiopharmaceuticals administered within 8 weeks prior to the first dose of study treatment; ≥ 3 weeks since the last chemotherapy or approved targeted therapy; biological therapy, immunotherapy, and other treatments must be completed at least 4 weeks prior to the first dose of study treatment.
5. ECOG performance status (Appendix 1) ≤ 2;
6. Expected survival > 12 weeks;
7. Hematological parameters must meet the following criteria: a) Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L; b) Hemoglobin (HGB) ≥ 80 g/L; c) Platelet count (PLT) ≥ 75 × 10^9/L, with no platelet or red blood cell transfusions within 2 weeks prior to screening. Note: If the investigator believes that the patient's laboratory values below the protocol limits are due to bone marrow involvement by lymphoma, the patient's eligibility may be determined after discussion with the sponsor and CRO medical team.
8. Liver and kidney function test results must meet the following criteria: a) Serum total bilirubin (TBiL) ≤ 1.5 × upper limit of normal (ULN); b) Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 × ULN; c) Serum creatinine ≤ 1.5 × ULN. Note: Patients with Gilbert's syndrome may be enrolled if TBiL ≤ 3.0 × ULN; patients with liver involvement by lymphoma may be enrolled if AST, ALT, and ALP ≤ 5 × ULN.
9. Left ventricular ejection fraction (LVEF) ≥ 50% as measured by echocardiography;
10. Women of childbearing potential and men must agree to use effective contraception from the time of signing the informed consent form until 6 months after the last dose of pomalidomide mesylate. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose. Women of childbearing potential include premenopausal women and women within 1 year of menopause.
11. Participants must voluntarily sign the informed consent form, be able to communicate effectively with the investigator, and comply with the study visit schedule, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria

1. Subjects who meet any of the following criteria will be excluded from the trial:
2. Known severe allergy to the investigational drug or any of its excipients;
3. Primary central nervous system lymphoma or lymphoma involving the central nervous system;
4. Prior chronic lymphoma transformation (e.g., Richter syndrome, prolymphocytic leukemia, etc.);
5. Presence of other active malignancies requiring treatment that may interfere with the study;
6. History of solid organ or allogeneic hematopoietic stem cell transplantation;
7. Coagulation abnormalities, defined as: international normalized ratio (INR) > 1.5 × upper limit of normal (ULN), prothrombin time (PT) > 1.5 × ULN, activated partial thromboplastin time (APTT) > 1.5 × ULN, thrombin time (TT) > 1.5 × ULN, or fibrinogen (FIB) < 1 g/L;
8. Active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV), except for the following:

   1. HBV infection: If hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) is positive, peripheral blood HBV DNA titer must be ≤ 1 × 10^3 copies/mL for enrollment; antiviral therapy must be continued after enrollment, and HBV DNA titer must be monitored every cycle;
   2. HCV seropositivity with negative HCV RNA test results is allowed for enrollment; Positive human immunodeficiency virus antibody (HIV-Ab) or positive syphilis antibody (TP-Ab) (patients with positive syphilis antibody in phase IIb may undergo titer testing, and eligibility will be determined by the investigator based on comprehensive assessment);
9. Any of the following cardiac function-related criteria:

   1. Clinically significant arrhythmias or conduction abnormalities requiring clinical intervention;
   2. Average corrected QT interval (QTcF) > 450 msec (male) or > 470 msec (female) based on three electrocardiogram (ECG) measurements (retesting is required only if the first ECG shows QTcF > 450 msec (male) or > 470 msec (female), and the average of three measurements will be used);
   3. History of long QT syndrome or confirmed family history of long QT syndrome; history of clinically significant ventricular arrhythmias, or current use of antiarrhythmic drugs or implanted defibrillator for ventricular arrhythmias;
   4. Clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina, coronary artery bypass grafting, or cardiomyopathy within 6 months prior to the first dose; congestive heart failure classified as New York Heart Association (NYHA) class 3 or higher, or left ventricular ejection fraction (LVEF) < 50%;
10. Other systemic diseases:

    1. Poorly controlled diabetes;
    2. Severe pulmonary disease (CTCAE V5.0 grade III-IV);
    3. History of psychiatric disorders, family history of psychiatric disorders, or mood disorders as judged by the investigator or psychiatrist, including medical records of depressive episodes, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, suicide attempts or suicidal ideation, or homicidal thoughts (immediate risk of harm to others), or anxiety of grade 3 or higher;
11. Prior treatment conditions:

    1. Chimeric antigen receptor T-cell immunotherapy (CAR-T therapy) within 3 months prior to the first dose;
    2. Prior treatment with HDAC inhibitors (except for chidamide) or other small molecule targeted therapies;
    3. Autologous hematopoietic stem cell transplantation within 3 months prior to the first dose;
    4. Radiotherapy affecting the efficacy evaluation of this study or local radiotherapy affecting bone marrow function within 3 months prior to the first dose;
    5. Myelosuppressive chemotherapy, biological therapy, or targeted therapy within 4 weeks prior to the first dose;
    6. Major surgery (excluding tumor biopsy) within 4 weeks prior to the first dose, or if the patient has not recovered or the side effects of surgery have not stabilized;
    7. Treatment with hematopoietic growth factors (e.g., granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF]), recombinant IL-11, thrombopoietin, or TPO-R agonists within 2 weeks prior to the first dose. Note: Subjects who started erythropoietin or darbepoetin treatment within 2 weeks prior to the first dose are eligible;
    8. Treatment with prednisone > 10 mg daily (or equivalent doses of other glucocorticoids, see Appendix 2) within 7 days prior to the first dose. Note: If used for non-lymphoma conditions such as rheumatoid arthritis, polymyalgia rheumatica, adrenal insufficiency, or asthma, subjects may receive a stable dose of prednisone up to 10 mg daily (or equivalent doses of other glucocorticoids);
12. Persistent grade 2 or higher toxicities (CTCAE V5.0 criteria) from prior treatment (chemotherapy, biological therapy, or targeted therapy) that have not recovered to ≤ grade 1 at the time of enrollment (excluding alopecia);
13. Uncontrolled active clinical infections of grade 2 or higher (CTCAE V5.0 criteria) requiring systemic anti-infective therapy (except if the infection is controlled but maintenance anti-infective therapy is still required);
14. Treatment within 7 days prior to the first dose with: known strong CYP3A4 inhibitors/inducers or drugs known to significantly prolong the QT interval (concomitant use of weak CYP3A4 inhibitors is allowed; see Appendix 3 for a list of common CYP3A4 inhibitors or inducers);
15. Participation in other interventional clinical trials within 4 weeks prior to the first dose;
16. Pregnant or breastfeeding women;
17. Alcohol or drug abusers;
18. Conditions that, in the investigator's judgment, may compromise the subject's safety or compliance;
19. Subjects deemed unsuitable for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of PM | each cycle lasts 21 days, and patients are assessed every 2 cycles until maximum of 2 years.
  proportion of patients whose tumors have shrunk to the pre-specified value and maintained for required minimum time，including CR and PR.

SECONDARY OUTCOMES:
TTR | each cycle lasts 21 days, and patients are assessed every 2 cycles until maximum of 2 years.
  The time between the first treatment and the first objective response
Duration of relief (DOR) of PM | each cycle lasts 21 days, and patients are assessed every 2 cycles until maximum of 2 years.
  The time from the first documentation of complete remission (CR) or partial remission (PR) to the first documentation of disease progression (PD)
Overall survival (OS) of PM | each cycle lasts 21 days, and patients are assessed every 2 cycles until maximum of 2 years.
  Time from the patient's first administration of Purinostat Mesylate for Injection to death from any cause.
Progression-free survival (PFS) of PM | each cycle lasts 21 days, and patients are assessed every 2 cycles until maximum of 2 years.
  Time from the patient's first administration of Purinostat Mesylate for Injection to the occurrence of disease progression (PD) or death, whichever occurs first.
Disease control rate (DCR) of PM | each cycle lasts 21 days, and patients are assessed every 2 cycles until maximum of 2 years.
  proportion of patients whose tumors have shrunk or remained stable for a certain period of time, including CR, PR and SD (stable disease) cases

CONTACTS AND LOCATIONS:
Overall Officials: Ting Niu, Doctor, Principal Investigator — West China Hospital; Weili Zhao, Doctor, Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Ruijin Hospital of Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No